CLINICAL TRIAL: NCT03338465
Title: Extracorporeal Shockwave Treatment in the Greater Trochanteric Pain Syndrome. Multicenter, Randomized, Controlled Clinical Trial
Brief Title: Extracorporeal Shockwave Treatment for Greater Trochanteric Pain Syndrome
Acronym: ESTATE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Maria Chiara Vulpiani, Head of Physical Medicine and Rehabilitation Unit, Sant'Andrea Hospital of Rome, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4
Record Dates: First submitted 2017-11-02; First posted 2017-11-09 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Mobility Limitation; Trochanteric Syndrome; Gluteal Tendinitis; Bursitis Hip; Pain Syndrome
Keywords: Greater Trochanteric Pain Syndrome,; Gluteal; Tendinopathy; ESWT; shockwave
MeSH Terms: conditions — Mobility Limitation; Somatoform Disorders; Tendinopathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants will be blinded to the type of ESWT treatment and the assessor, data managers, statistician and study monitors will be blinded to the allocation. All participants who receive ESWT treatment will be treated using the same device (Duolith SD1, STORZ Medical, Switzerland) regardless of what group they are included in. The participants will not be able to predict the allocated group based on the appearance of the ESWT treatment. The blinding will be maintained until the data are locked. For blinding evaluation, allocation guessing will be assessed immediately after the final treatment. Practitioners and assessors will be instructed to treat the participants according to predefined standard operating procedures during the trial to maintain blinding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A (Active Comparator): 3 weekly sessions of focused extracorporeal shockwave treatment (2.000 impulses at 0.20 millijoules/mm2 per session)
  Interventions: Device: Duolith SD1, STORZ Medical, Switzerland with F-SW applicator
- Group B (Active Comparator): 3 weekly sessions of focused extracorporeal shockwave treatment (2.000 impulses at 0.01 millijoules/mm2 per session)
  Interventions: Device: Duolith SD1, STORZ Medical, Switzerland with F-SW applicator

INTERVENTIONS:
Device: Duolith SD1, STORZ Medical, Switzerland with F-SW applicator — The procedure will be performed with the patient in lateral positioning of the decubitus. The treatment area will be prepared with a coupling ultrasound gel to minimize the loss of shockwave energy at the interface between the tip of the applicator and the skin. The inline ultrasonic guide will be used to concentrate the shockwaves on the pain area in the trochanteric region. No local anesthesia will be applied.
  Other Names: Focused Extracorporeal Shock Waves; ESWT

SUMMARY:
Greater trochanteric pain syndrome (GTPS) is characterized by pain over the greater trochanter, which can refer down the lateral aspect of the hip. Historically, conservative treatments such as rest/activity modification, anti-inflammatory medication, physiotherapy and local corticosteroid injection, are employed as first-line management, with some refractory cases requiring surgical intervention.

Acknowledging the unpredictable response and frequent recurrences associated with traditional non operative treatment, the risks and prolonged rehabilitation associated with surgery, and the favorable results from prior studies involving radial pressure waves as a treatment for GTPS, the aim of this study is to investigate the dose-related effect of focalized shockwave treatment at different total energy influx in patients with chronic GTPS.

DETAILED DESCRIPTION:
Shockwave therapy (SWT) has been used successfully since the late 1980s for the management of various musculoskeletal disorders including plantar fasciopathy, achilles tendinopathy, shoulder calcific tendinopathy, and lateral epicondylitis. Although there are some negative trials, there are now many randomized, double-blinded, clinical trials that support the use of SWT for the above conditions. Acknowledging the unpredictable response and frequent recurrences associated with traditional non operative treatment, the risks and prolonged rehabilitation associated with surgery, the recognition of gluteal tendinopathy as a potential source of pain, and the favorable results from prior studies involving radial pressure waves as a treatment for GTPS, the aim of this study is to investigate the dose-related effect of shockwave treatment at different total energy by adjusting the energy flux density (EFD) in patients with chronic GTPS. The shockwave has been widely recognized in literature as a biological regulator, currently the biological effects of shockwaves can be obtained using lower energy than in the past.

While the intensity or delivered energy is considered by some researchers to be a key factor for successful treatment, in current literature reviews, debate continues over the appropriate energy intensity and the total delivered energy that should be applied to the tissue.

Therefore, higher intensity treatments usually require local anesthesia, which is known to reduce the efficacy of the treatment. Furthermore, some animal tests reported that an influx of energy of over 0.60 mJ/mm2 can cause permanent damage on the tendon. On the other hand, low-intensity energy is safer but has the disadvantage of lower treatment effects.

The investigators hypothesize that a very low intensity protocol of ESWT has different effects on pain and function than a conventional protocol in a patient with GTPS syndrome.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of either sex, aged oved 18 years, complaining of pain located anterior, lateral or posterior to the great trochanter for more than 3 months.
2. Pain while lying on the affected side.
3. Local tenderness on palpation of the area of the great trochanter of patients with this symptom as the reason for the consultation.

Exclusion Criteria:

1. Presence of signs and symptoms of another cause of regional hip pain.
2. Presence of hip internal rotation 20° and extension deficit or other range of motion limitation 10º
3. Previous hip surgery or use of ESWT for GTPS.
4. Acute low back pain
5. Vascular, neurologic, rheumatic diseases.
6. Tumor in the area or local infection to the hip joint region.
7. Pregnancy.
8. Severe coagulation disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) for the estimation of the intensity of pain | 8 weeks after treatment (T2)
  The VAS provides a continuous scale for magnitude estimation and consists of a straight line, the ends of which are defined in terms of the extreme limits of pain experience such as 'no pain at all' and 'pain as bad as it could be'. Respondents mark the location on the 10-centimeter line corresponding to the amount of pain experienced. This gives the greatest freedom to choose pain's exact intensity. It also gives the maximum opportunity for each respondent to express a personal response style. VAS data of this type is recorded as the number of millimeters from the left of the line with the range 0-100.

SECONDARY OUTCOMES:
Harris Hip Score (HHS) to evaluate hip disability | 4 (T1), 8 (T2), 12 (T3) and 24 (T4) weeks after treatment.
  The index consists of questions about pain and activities of daily living, referring to the previous week, and assessments of hip function (limping) and range of motion. Score ranges from 100 (no disability) to 0 (maximum disability).
Lower Extremity Functional Scale (LEFS) | 4 (T1), 8 (T2), 12 (T3) and 24 (T4) weeks after treatment.
  The LEFS is a self-report questionnaire to measure "patients' initial function, ongoing progress, and outcome about Lower Extremity. Patients will answer the question "Today, do you or would you have any difficulty at all with:" in regards to twenty different everyday activities. The maximum possible score is 80 points, indicating very high function. The minimum possible score is 0 points, indicating very low function.
Roles and Maudsley scale (RM) to evaluate patients satisfaction | 4 (T1), 8 (T2), 12 (T3) and 24 (T4) weeks after treatment.
  The RM scale is a subjective 4-point patient assessment of pain and limitations of activity. The RM score has been used extensively at centers throughout the world to assess outcome after SWT. On the scale, 1 point indicates an excellent result with the patient having no symptoms. Two points indicate a good result with the patient significantly improved from the pretreatment condition and satisfied with the result. Three points indicate a fair result with the patient somewhat improved from the pretreatment condition and partially satisfied with the treatment outcome. Four points indicate a poor outcome with symptoms identical or worse than the pretreatment condition and dissatisfaction with the treatment result.
EuroQoL five dimensions questionnaire (EQ-5D) to evaluate quality of life | 4 (T1), 8 (T2), 12 (T3) and 24 (T4) weeks after treatment.
  The EQ-5D consists of two distinct sections.The first one is a subjective assessment for five dimensions (mobility, self-care, daily activities, pain / discomfort and anxiety / depression) and each item provides the option to choose a level of gravity. Each item provides graduated answers from 1 to 3. The Level 1 is no problem, while leveling 3 the extreme limitation. The aggregation of the responses forms a five-digit number that represents the state of health. The three levels of response, for each of the five items, produce up to 243 possible descriptions of the state of health and allow to highlight the presence / absence of any problems and the their intensity.
  The second section of the EQ-5D includes a VAS scale, represented graphically from a graduated scale ranging from 0 (worst possible health) at 100 (the best possible state of health) on which the interview indicates his perceived level of health status.
Visual Analogue Scale (VAS) for the estimation of the intensity of pain | 4 (T1), 12 (T3) and 24 (T4) weeks after treatment.
  The VAS provides a continuous scale for magnitude estimation and consists of a straight line, the ends of which are defined in terms of the extreme limits of pain experience such as 'no pain at all' and 'pain as bad as it could be'. Respondents mark the location on the 10-centimeter line corresponding to the amount of pain experienced. This gives the greatest freedom to choose pain's exact intensity. It also gives the maximum opportunity for each respondent to express a personal response style. VAS data of this type is recorded as the number of millimeters from the left of the line with the range 0-100.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Chiara Vulpiani, MD, PHD, Principal Investigator — Università Sapienza Roma
Locations (1):
- Sant'Andrea Hospital, Roma, RM, Italy